CLINICAL TRIAL: NCT00133406
Title: Long-term Impact and Intervention for Diarrhea in Brazil
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Richard Guerrant, University of VA
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12475; 05-0071 (Other: NIAID); NCT00421382 (obsolete NCT alias)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Diarrheal Disorder
Keywords: Brazil, Child Nutrition Disorders, Deficiency Diseases
MeSH Terms: conditions — Child Nutrition Disorders; Deficiency Diseases | interventions — Glutamine; Vitamin A; Glycine; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- a (Experimental): oral glutamine with juice for 10 days
  Interventions: Drug: Glutamine
- b (Experimental): PO vit A q 4 mo for 1 year plus zinc placebo
  Interventions: Drug: Vitamin A; Drug: zinc
- c (Active Comparator): Zinc 40 mg twice weekly Plus Vitamin A Placebo for one year
  Interventions: Drug: Vitamin A; Drug: zinc
- d (Placebo Comparator): oral glycine with juice daily for 10 days
  Interventions: Drug: glycine
- e (Placebo Comparator): Vitamin A Placebo plus Zinc Placebo for one year
  Interventions: Drug: Vitamin A; Drug: zinc
- f (Experimental): Vitamin A q 4 months and PO Zinc for 1 year
  Interventions: Drug: Vitamin A; Drug: zinc

INTERVENTIONS:
Drug: Glutamine — 0.8gm/kg, ie up to a total daily dose of 16.2gm/day,with juice daily for 10 days
  Arms: a
Drug: Vitamin A — 100,000 IU for children under 12 months of age (or placebo) and PO 200,000 IU for children at least 12 months of age (or placebo), both q months for 1 year at 0, 4 and 8 months.
  Arms: b; c; e; f
Drug: glycine — 0.4gm/kg; ie up to 8.3gm/d, with juice daily for 10 days
  Arms: d
Drug: zinc — 40 mg twice weekly for 12 months
  Arms: b; c; e; f

SUMMARY:
The primary objectives of this study are to determine the effect of 1 year supplementation of Vitamin A, Zinc, and Vitamin A plus Zinc compared to placebo on the Height for Age Z Score (HAZ) and the number of episodes of diarrhea and number of days of diarrhea at one year in children living in a Brazilian slum. Study participants will include 280 children ages 2 months to 8 years old, with a Height for Age Z score (HAZ) less than median for the Parque Universitario community, living in Brazilian favela. There is also a sub study to determine if ten days of glutamine delivered as an oral bolus improves the health of the digestive system.

DETAILED DESCRIPTION:
Study participants will include 280 children ages 2 months to 8 years old, with a Height for Age Z score (HAZ) less than median for the Parque Universitario community, living in Brazilian favela. Subjects will be enrolled into this prospective, randomized, placebo controlled study of the Long-term Impact and Intervention for Diarrhea in Brazil. Children meeting the inclusion criteria will be prospectively, randomized to four arms: (1) placebo: placebo (2) Vitamin A: Zinc Placebo (3) Vitamin A Placebo:Zinc (4) Vitamin A:Zinc. Intervention will last for one year with two additional years of follow up. A nested study involving all patients will take place at week four. At week four there will be a second randomization to either oral glutamine or glycine (placebo) for an additional ten days. The primary endpoint of the nested study will be the L:M ratio at 6 weeks. The master randomization list will be broken, only by combined approval of the Principal Investigators, at the end of the study or in the unexpected event of a child needing removal from the study (for that case only). All randomized subjects will be visited in their home two times per week for assessment of intercurrent diarrhea. At 1, 4, 8, 12, 24 and 36 months patients will have a nutritional status/anthropometry and diarrheal illness rate assessment. At 0, 1, 1.5, and 4 months all randomized subjects will have a Lactulose:Mannose Ratio (L:M) performed. A blood Zinc and Vitamin A level will be drawn at 0 and 4 months. Also a stool microbiology, lactoferrin and protein loss assessment will be completed at 1 month. All randomized subjects who complete the protocol should have assessments as outlined above at 36 weeks. The primary effect of interest is the difference in mean HAZ changes between children receiving Zinc plus Vitamin A compared to children receiving no Vitamin A or Zinc, averaging the difference in children receiving glutamine and children not receiving glutamine.

ELIGIBILITY:
Inclusion Criteria:

Children ages 2 months to 8 years with height for age Z-score (HAZ) less than the median for the Parque Universitario community. Be a resident in Brazilian flavela. Child's parent or guardian must sign informed consent.

Exclusion Criteria:

Children exclusively breast-fed. Children who participated in the "hospital study" or any other study with in the past two years. Children with fever > 102 F at time of screening. Children with systemic disease at the time of screening including but not limited to: shock, meningitis, sepsis, pneumonia, tuberculosis, varicella. Children on antibiotics during screening. Children with siblings from the same household enrolled in this study.

Ages: 2 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 321 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
L:M ratio at 1.5 months | 1.5 months

SECONDARY OUTCOMES:
L:M ratio at 4 & 12 months | 4 and 12 months
HAZ | 1.5, 4, 8, 12, 24, and 36 months
Diarrhea burden | 4, 8, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Guerrant, MD, Principal Investigator — University of Virginia
Locations (1):
- Federal University of Ceará, Fortaleza, Brazil

REFERENCES:
- [Derived] Lima AA, Anstead GM, Zhang Q, Figueiredo IL, Soares AM, Mota RM, Lima NL, Guerrant RL, Oria RB. Effects of glutamine alone or in combination with zinc and vitamin A on growth, intestinal barrier function, stress and satiety-related hormones in Brazilian shantytown children. Clinics (Sao Paulo). 2014;69(4):225-33. doi: 10.6061/clinics/2014(04)02. PMID 24714829
- [Derived] Lima AA, Kvalsund MP, Souza PP, Figueiredo IL, Soares AM, Mota RM, Lima NL, Pinkerton RC, Patrick PP, Guerrant RL, Oria RB. Zinc, vitamin A, and glutamine supplementation in Brazilian shantytown children at risk for diarrhea results in sex-specific improvements in verbal learning. Clinics (Sao Paulo). 2013;68(3):351-8. doi: 10.6061/clinics/2013(03)oa11. PMID 23644855
- [Derived] Mitter SS, Oria RB, Kvalsund MP, Pamplona P, Joventino ES, Mota RM, Goncalves DC, Patrick PD, Guerrant RL, Lima AA. Apolipoprotein E4 influences growth and cognitive responses to micronutrient supplementation in shantytown children from northeast Brazil. Clinics (Sao Paulo). 2012;67(1):11-8. doi: 10.6061/clinics/2012(01)03. PMID 22249475
- [Derived] Lima AA, Soares AM, Lima NL, Mota RM, Maciel BL, Kvalsund MP, Barrett LJ, Fitzgerald RP, Blaner WS, Guerrant RL. Effects of vitamin A supplementation on intestinal barrier function, growth, total parasitic, and specific Giardia spp infections in Brazilian children: a prospective randomized, double-blind, placebo-controlled trial. J Pediatr Gastroenterol Nutr. 2010 Mar;50(3):309-15. doi: 10.1097/MPG.0b013e3181a96489. PMID 20038852